CLINICAL TRIAL: NCT04392713
Title: Efficacy of Ivermectin in COVID-19 : A Randomized Controlled Trial
Brief Title: Efficacy of Ivermectin in COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Asma Asghar, Consultant Medicine, Combined Military Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVE-COV
Record Dates: First submitted 2020-05-05; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: COVID
MeSH Terms: interventions — Ivermectin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin arm (Active Comparator): Participants will be administered Ivermectin with standard chloroquine regimen
  Interventions: Drug: Ivermectin 6 MG Oral Tablet (2 tablets)
- Control arm (No Intervention): This arm will only receive chloroquine as per existing policy of hospital

INTERVENTIONS:
Drug: Ivermectin 6 MG Oral Tablet (2 tablets) — 12 mg single dose of Ivermectin will be given to intervention arm
  Arms: Ivermectin arm

SUMMARY:
It is a randomized controlled trial to assess the efficacy of Ivermectin in COVID-19. Patient recruited will be assigned to two groups one group will be given ivermectin with standard chloroquine regimen and the other group will be receiving chloroquine only. Out come will be recorded by documenting PCR reports at 48, 96 and 144 hours.

DETAILED DESCRIPTION:
INTERVENTION It will be a randomized controlled trial which will be done on COVID-19 patients proven by PCR fulfilling the criteria (asymptomatic/mild to moderate severity). They will be divided into two groups after randomization. Group A will be administered Ivermectin single dose of 12grams along with Chloroquine as per existing hospital guidelines and group B will be given Chloroquine alone. Dose of Ivermectin to be repeated at 1 week if PCR stays negative. PCR will be done on alternate days (48, 96 and 144hours) and the duration at which the PCR becomes negative will be compared. Dose of drug subject to change in accordance with patient response or possible side effect.

ELIGIBILITY CRITERIA INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Provision of signed and dated informed consent form Stated willingness to comply with all study procedures and availability for the duration of the study Male or female, aged 15 to 65 years In good general health with no or mild symptoms of Corona virus disease PCR positive for SARS-Cov-2. Ability to take oral medication and be willing to adhere to the drug intake regimen EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

Severe symptoms likely attributed to Cytokine Release Storm. Malignant diseases, diabetes mellitus, chronic kidney disease and cirrhosis liver with CPT class B or C.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 15 to 65 years
* In good general health with no or mild to moderate symptoms of Corona virus disease
* PCR positive for SARS-Cov-2.
* Ability to take oral medication and be willing to adhere to the drug intake regimen

Exclusion Criteria:

* Severe symptoms likely attributed to Cytokine Release Storm.
* Malignant diseases, diabetes mellitus, chronic kidney disease and cirrhosis liver with CPT class B or C.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Negative PCR | 144 hours
  PCR will be done at 48, 96 and 144 hours

SECONDARY OUTCOMES:
Need for mechanical ventilation | 4 weeks
  All patients will be assessed for requirement of mechanical ventilation in both the groups

CONTACTS AND LOCATIONS:
Overall Officials: Karamat Hu Bukhari, FCPS MED, Study Director — Combined military hospital lahore
Locations (1):
- Combined Military Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Result] Simsek Yavuz S, Unal S. Antiviral treatment of COVID-19. Turk J Med Sci. 2020 Apr 21;50(SI-1):611-619. doi: 10.3906/sag-2004-145. PMID 32293834